CLINICAL TRIAL: NCT04979858
Title: Reducing Spread of COVID-19 in a University Community Setting: Role of a Low-Cost Reusable Form-Fitting Fabric Mask for Community Use
Brief Title: Reducing Spread of COVID-19 in a University Community Setting: Role of a Low-Cost Reusable Form-Fitting Fabric Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H21218; 75D30121C10545 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2021-07-22; First posted 2021-07-28 (Actual); Results first posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Covid19; SARS-CoV2 Infection
Keywords: Reusable masks; University Setting
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: One group will receive the focal mask and the other group will choose its own mask.
Who Masked: Investigator
Masking Description: The PI will not know which subjects have been assigned to which arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control Group (No Intervention): The subjects will choose their own mask and masking practices.
- Treatment Group (Experimental): The treatment group will receive and use the focal mask.
  Interventions: Device: Focal Mask

INTERVENTIONS:
Device: Focal Mask — The treatment group will receive and use the focal mask.
  Arms: Treatment Group

SUMMARY:
The primary aim of the proposed research is to test the role of a newly developed reusable form-fitting fabric mask in reducing the spread of COVID-19 in a community setting comprising undergraduate students living in dormitories at the Georgia Institute of Technology (Georgia Tech). A corollary aim is to assess the role of wearing any type of face covering in reducing spread in the same community setting. A final aim is to assess the social, behavioral, aesthetic, and usability aspects of wearing face coverings in public settings.

DETAILED DESCRIPTION:
The primary aim of the proposed research is to test the role of a newly developed reusable form-fitting fabric mask in reducing the spread of COVID-19 in a community setting comprising undergraduate students living in dormitories at Georgia Tech. The study has been designed such that it also leads to the corollary aim of assessing the role of wearing any type of face covering in reducing spread in the same community setting. Yet another aim is to assess the social, behavioral, aesthetic, and usability aspects of wearing face coverings in public settings. The study design is to assign student users of masks randomly to the Treatment group of focal mask users (n=100) and a Control group of other mask users (n=100).

The Study Population and Data Collection: The subject population will comprise 200 undergraduate students staying in the dormitories at Georgia Tech, preferably freshmen and sophomores with meal plans. There will be no restriction of race, gender, or sexual orientation for this study. The final cohort chosen will attempt to reflect the demographics of the undergraduate student body at Georgia Tech. The participating subjects will have the option to withdraw from the study at any time. The recruitment of subjects will be carried out in collaboration with Georgia Tech Housing through e-mail and web announcements. The research team will be accessible to the subjects at all times during the study.

As part of the informed consent process during recruitment, the Treatment Group will be told about the use, care and laundering of the focal mask during the study. The planned sample size of 200 accounts for dropouts, which are likely to occur so that a statistically significant sample is present to assess the effect of the mask. A randomized study cannot be undertaken for ethical and practical reasons (e.g., the fact that the behaviors of students cannot be controlled leading to heterogeneity); therefore, a DID (Difference-in-Difference) approach that has been used extensively in public health research will be utilized in this study . The DID method assumes that unobserved heterogeneity in participation is present but that such factors are time invariant. With data on observations before and after the treatment intervention, this fixed component can be differenced out. For this reason, the study is spread over six weeks consisting of three phases: Pre-treatment, Treatment, and Post-treatment, with each phase lasting two weeks. The two-week period for each phase is based on the following rationale: The incubation period of COVID-19 virus has been found to be five days. About 97% of the people who get infected and develop symptoms will do so within 11 to 12 days, and about 99% will within 14 days, which is the basis for the 14-day quarantine recommended by Centers of Disease Control. The health and well-being of the subjects will be tracked during the study. Any student falling sick will be given medical help using on-campus health services. Georgia Tech has a system in place with the ability to conduct 1,500 tests per day, going to possibly 3,000 per day. If the COVID-19 test is positive, the subject will be excluded from the remainder of the study. The subject will, however, be compensated at the end of the study.

Data Collection: During the study, demographic, behavioral, and mask use data will be recorded and appropriately de-identified. No specimens will be obtained from the subjects. All the collected data will be access limited, and destroyed when no longer needed to perform the study or analysis or after completion and publication of the study, whichever comes first. COVID-19 diagnoses will be self-reported by the subjects.

At the beginning of the study, each subject will provide the following data:

* Subject Profile: Demographic information, class schedule, dining plans
* Baseline Practice Data: Mask usage practice (type, duration), typical social interactions
* During the study, each subject will provide the following data every day:
* Health Metrics: Temperature, Typical COVID-19 symptoms (if any)
* Mask Usage Data: Type and duration of mask usage including washing
* Activity Data: Classes attended, group meetings, social and dining interactions

At the end of the study, each subject will provide the following data:

* Usability: Comfort, Ease of Donning/Doffing, Impact on Communication
* Shape Conformability: Conforms to face, Shape retention after washing
* Ease of Care: Ease of washing
* Aesthetic and Social Perceptions: Style, Perceptions of others, Impact on personal behavior and degree of social interactions

The Difference-in-Difference (DID) methodology will be used to analyze the data from the Control and Treatment groups. The difference in infection rates between the groups will help determine the role of the focal mask.

ELIGIBILITY:
Inclusion Criteria:

* Georgia Institute of Technology (Georgia Tech) student
* 18 years old or older
* Living on campus in Georgia Tech dorms

Exclusion Criteria:

* Not a Georgia Tech student
* Under the age of 18
* Not living on campus in Georgia Tech dorms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundaresan Jayaraman, Ph.D, Principal Investigator — Georgia Institute of Technology
Locations (1):
- Georgia Institute of Technology - Main Campus, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Pre-Treatment
Arm/Group | Control Group | Treatment Group
Started (At the beginning of the study, 201 participants were enrolled. One of the participants was in "quarantine" at that time. Additionally, during Pre-Treatment, all participants were considered to be in the Control Group. After Pre-Treatment, the participants were randomly assigned to either remain in the Control Group or be assigned to the Treatment Group.) | 201 | 0
Completed (The participant who had been quarantining developed contracted COVID-19 and withdrew from the Study in accordance with the Study Protocol. Hence the number at the end of the Pre-Treatment phase was 200.) | 200 | 0
Not Completed | 1 | 0
Not completed — The participant was in quarantine at start of study and contracted COVID-19. | 1 | 0
Period: Treatment
Arm/Group | Control Group | Treatment Group
Started (The participant who contracted COVID-19 in the Pre-Treatment phase withdrew from the study in accordance with the Study Protocol.) | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0
Period: Post-Treatment
Arm/Group | Control Group | Treatment Group
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Treatment Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Median (Full Range); unit: years] | 18 [18 to 22] | 18 [18 to 22] | 18 [18 to 22]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 49 | 49 | 98
  Female | 50 | 47 | 97
  Prefer Not to Say | 1 | 1 | 2
  Non-binary | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 90 | 93 | 183
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 56 | 48 | 104
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 30 | 41 | 71
  More than one race | 11 | 8 | 19
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Infected by COVID-19
Description: Number of participants not infected by COVID-19 in a university setting.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Treatment Group
Number analyzed (Participants) | 100 | 100
Participants | 100 | 100
Statistical Analysis 1: Comparison: Control Group vs Treatment Group; Test type: Other — The statistical analysis involved the use of a single-factor ANOVA test to assess the importance of the various factors associated with the design of the Focal Mask (the Treatment) that would impact its performance in reducing the spread of COVID-19, which is caused by the SARS-CoV-2 virus. The Bonferroni t-test was conducted post hoc to assess the statistical significance of the various factors; p < 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: Six weeks.
Description: Same as clinicaltrials.gov
Arm/Group | Control Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

LIMITATIONS AND CAVEATS:
To simulate a "real" community setting in which individual behaviors cannot be specified, monitored, or controlled, regular health diagnostic testing for COVID-19 during the study was not mandated for the subjects. Therefore, subjects who became infected, but were asymptomatic, would not have been tested; as a result, there is a potential for undercounting the number of reported positive cases during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04979858/Prot_001.pdf
  • Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04979858/SAP_002.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT04979858/ICF_000.pdf